CLINICAL TRIAL: NCT00601770
Title: Open-label, Multicenter Trial With IC41, a Therapeutic HCV Vaccine in Patients With Chronic HCV
Brief Title: Virological Response Study of the HCV Vaccine IC41
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC41-202
Record Dates: First submitted 2008-01-04; First posted 2008-01-28 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IC41 (Experimental): 8 injections of 4 x 0.125mL
  Interventions: Biological: IC41

INTERVENTIONS:
Biological: IC41 — injection

SUMMARY:
The objective is to investigate the virological (HCV-RNA) responses following biweekly immunization with IC41.

Treatment phase 14 weeks, total study duration including follow-up period 38 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to study entry
* Patients with chronic hepatitis C; genotype 1
* Treatment naive patients
* Male and Female, 18 to 55 years
* Presence of HLA-A2 marker
* Mentally healthy
* No clinically relevant pathological findings in any of the investigations at screening
* Treatment naive patients with chronic Hepatitis C of genotype 1

Exclusion Criteria:

* Positive results in HIV, HBsAg and HAV-Ag (IgM)
* Other causes of chronic hepatitis
* History of autoimmune diseases
* Previous vaccination with any prophylactic or therapeutic Hepatitis C vaccine (in a clinical study)
* Active or passive vaccination 4 weeks before and during the entire study period
* Decompensated liver disease
* History of severe hypersensitivity reactions and anaphylaxis
* Known allergic reactions to one of the components of the vaccine and Imiquimod cream
* Clinically significant diseases which, in the opinion of the Investigator, might lead to frequent hospitalization/medical attendance
* Malignancies
* Immunosuppressive therapy
* Pregnancy, lactation or breast-feeding
* Unwillingness to practice appropriate contraception
* Participation in another study with an investigational drug within 1 month prior to enrolment and the entire study period
* Patients, who in the opinion of the Investigator, might not be able to comply with the study protocol (e.g.: Drug addiction, alcoholism)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
HCV-RNA 2 weeks after end of treatment | 2 weeks

SECONDARY OUTCOMES:
Immunological assays and Safety | until study end

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Ernsthofer, Mag, Study Director — Valneva Austria GmbH
Locations (8):
- Germany (2):
  - Prof. Dr. Ulrich Spengler, Bonn, Bonn
  - Prof. Dr. Michael Manns, Hanover, Hannover
- Poland (2):
  - Dr. Granzyna Cholewinska-Szymanska, Warzawa, Warzawa
  - Prof. Dr. Andrzej Gladszy, Wroclaw, Wroclaw
- Romania (4):
  - Prof. Dr. Mircea Diculescu, Bucharest, Bucharest
  - Dr. Adriana Motoc, Bucharest, Bucharest
  - Dr. Adriana Hristea, Bucharest, Bucharest
  - Prof. Dr. Carol Stanciu, Iași, Iaşi